CLINICAL TRIAL: NCT03798509
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of Human CD19 Targeted T Cells Injection for Subjects With Relapsed and Refractory CD19-positive B-cell Acute Lymphoblastic Leukemia
Brief Title: Human CD19 Targeted T Cells Injection Therapy for Relapsed and Refractory CD19-positive Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-ALL01
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: CD19-positive; Acute Lymphoblastic Leukemia
Keywords: CD19; CAR-T; leukemia; Relapsed /Refractory; B-ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human CD19 targeted T Cells Injection (Experimental)
  Interventions: Drug: Human CD19 targeted T Cells Injection

INTERVENTIONS:
Drug: Human CD19 targeted T Cells Injection — Autologous genetically modified anti-CD19 CAR transduced T cells

SUMMARY:
To evaluate the safety and tolerance of human CD19 targeted T Cells injection for the treatment of relapsed and refractory CD19-positive B-cell acute lymphoblastic leukemia. Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19 CAR+ T cells.

DETAILED DESCRIPTION:
Participants with relapsed/refractory CD19-positive B-cell acute lymphoblastic leukemia can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, electrocardiograph and blood draws. Participants receive chemotherapy prior to the infusion of CD19 CAR+ T cells. After the infusion, participants will be followed for side effects and effect of CD19 CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 Years Old, Male and female;
2. Expected survival > 12 weeks;
3. ECOG score 0-1;
4. Bone marrow examination clearly diagnosed as CD19 positive B-cell acute lymphoblastic leukemia and who met one of the following conditions:

   1. Those who failed to achieve CR after at least 2 courses of standard chemotherapy or had early relapse after complete remission (<12 months) or late relapse after complete remission (≥ 12 months) and failed to achieve CR after 1 course of standard chemotherapy;
   2. For Ph+ ALL: in addition to receiving at least 2 courses of standard chemotherapy, at least two TKIs should be treated with no complete remission or relapse after complete remission (Patients who cannot tolerate TKI therapy or have TKI treatment contraindications or have T315i mutation are excluded);
   3. Those who relapse after stem cell transplantation are not affected by previous treatments;
5. The venous access required for collection can be established and mononuclear cell collection can be determined by the investigators;
6. Liver, kidney and cardiopulmonary functions meet the following requirements:

   1. Creatinine is in the normal range;
   2. Left ventricular ejection fraction >50%;
   3. Baseline oxygen saturation>92%;
   4. Total bilirubin ≤ 2×ULN; ALT and AST ≤2.5 × ULN;
7. Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

1. Graft-versus-host disease (GVHD), or need to use immunosuppressants;
2. Malignant tumors other than acute lymphoblastic leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
3. Subjects with positive HBsAg or HBcAb and peripheral blood HBV DNA titer detection ≥ 1 × 102 copy number / L; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; CMV DNA positive; syphilis positive;
4. Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
5. Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
6. Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
7. Received CAR-T treatment or other gene therapies before enrollment;
8. Patients with symptoms of central nervous system;
9. Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
10. The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days post infusion

SECONDARY OUTCOMES:
Duration of CAR-positive T cells in circulation | 2 years post infusion
The concentration of CD19-positive B cells in peripheral blood. | 2 years post infusion
Overall response rate (ORR) after administration | 90 days post infusion
Duration of remission (DOR) after administration | 2 years post infusion
Progress Free Survival (PFS) after administration | 2 years post infusion
Overall Survival (OS)after administration | 2 years post infusion
The immunogenicity of Human CD19 targeted T Cells Injection. (the detection of human anti-mouse antibody) | 2 years post infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Tsao ST, Gu M, Fu C, He F, Li X, Zhang M, Li N, Hu HM. A simple and effective method to purify and activate T cells for successful generation of chimeric antigen receptor T (CAR-T) cells from patients with high monocyte count. J Transl Med. 2022 Dec 19;20(1):608. doi: 10.1186/s12967-022-03833-6. PMID 36536403